CLINICAL TRIAL: NCT07280598
Title: Taking Advantage of Phage Technologies (TAPT) to Facilitate Phage Therapy While Reducing the Use of Antibiotics in the Management of Cystic Fibrosis (CF)
Brief Title: Safety of Combined Intravenous Antibiotic and Bacteriophage Therapy in Adults With Cystic Fibrosis and Antibiotic-Resistant Lung Infections
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, David Pride, Director of the Clinical Molecular Microbiology Laboratory, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 812895; 314645-00001 (Other Grant/Funding Number: Emily's Entourage); NCT07048704 (obsolete NCT alias)
Record Dates: First submitted 2025-11-20; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: CF - Cystic Fibrosis; Klebsiella Pneumoniae Infection; E Coli Infections; Staphylococcus Aureus Infection; Achromobacter; Stenotrophomonas Maltophilia Infection
Keywords: cystic fibrosis; CF; Phage; bacteriophage
MeSH Terms: conditions — Cystic Fibrosis; Escherichia coli Infections; Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 Study of Combined IV Antibiotics and Bacteriophage Therapy for Antibiotic-Res (Experimental): This arm will evaluate the safety and microbiological activity of a combined intravenous (IV) antibiotic and bacteriophage therapy in adults with cystic fibrosis (CF) who are experiencing pulmonary exacerbations caused by antibiotic-resistant bacterial pathogens. Participants will receive a clinician-selected, standard IV antibiotic regimen for 7 days, administered twice daily. In parallel, participants will receive a matched, pathogen-specific bacteriophage cocktail via IV infusion, also administered twice daily for 7 days. The phage cocktails consist of four lytic bacteriophages targeting one of the following pathogens: Pseudomonas aeruginosa, Klebsiella spp., Stenotrophomonas maltophilia, Escherichia coli, Staphylococcus aureus, or Achromobacter xylosoxidans. The first three phage doses will be administered in a monitored clinic setting; remaining doses will be self-administered at home via PICC line. This is a Phase 1, open-label, multi-site pilot study focused on safety.
  Interventions: Drug: Intravenous Bacteriophage Cocktail plus Standard IV Antibiotics

INTERVENTIONS:
Drug: Intravenous Bacteriophage Cocktail plus Standard IV Antibiotics — Participants will receive a seven-day course of intravenous (IV) bacteriophage therapy in combination with standard IV antibiotics. The bacteriophage therapy consists of a pathogen-specific cocktail containing four purified, lytic bacteriophages selected based on pre-treatment sensitivity testing of the participant's bacterial isolate. Each phage cocktail targets one of the following antibiotic-resistant pathogens: Pseudomonas aeruginosa, Klebsiella spp., Stenotrophomonas maltophilia, Escherichia coli, Staphylococcus aureus, or Achromobacter xylosoxidans. Phage cocktails are administered IV twice daily at a concentration of 1x10⁹ PFU/mL, following antibiotic infusion. The first three doses are observed in clinic; remaining doses are self-administered at home via PICC line. All phages are produced under GMP conditions and screened to be lytic-only, free of known toxin, resistance, or lysogeny genes.

SUMMARY:
This is a Phase 1, open-label, multi-center pilot study evaluating the safety and microbiological activity of intravenous (IV) bacteriophage therapy in combination with standard IV antibiotics in adults with cystic fibrosis (CF) experiencing pulmonary exacerbations due to antibiotic-resistant bacterial infections. Eligible participants will receive a 7-day course of IV antibiotics, selected by their treating clinician, along with a phage cocktail specifically formulated to target their identified bacterial pathogen (Pseudomonas aeruginosa, Klebsiella spp., Stenotrophomonas maltophilia, Escherichia coli, Staphylococcus aureus, or Achromobacter xylosoxidans). The primary objective is to assess the safety and tolerability of this combined treatment approach. Secondary and exploratory outcomes include assessment of changes in sputum bacterial burden, lung function (spirometry and oscillometry), quality of life, and bacteriophage pharmacokinetics. Results from this study will inform the feasibility and design of future clinical trials using phage therapy in the CF population.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a genetic disease characterized by chronic and recurrent pulmonary infections, often caused by antibiotic-resistant bacteria. These infections contribute significantly to lung function decline, reduced quality of life, and early mortality. Given the rising prevalence of antimicrobial resistance (AMR) and limited efficacy of conventional antibiotic therapies, there is an urgent need for novel therapeutic strategies. Bacteriophage (phage) therapy-using viruses that infect and lyse specific bacteria-has emerged as a promising, targeted approach for managing drug-resistant bacterial infections.

This is a Phase 1, open-label, multi-center pilot study designed to assess the safety, tolerability, and preliminary biological activity of intravenous (IV) bacteriophage therapy administered in combination with standard IV antibiotics in adults with CF experiencing a pulmonary exacerbation caused by antibiotic-resistant bacterial pathogens. Participants must have a confirmed diagnosis of CF and recent culture-proven infection with one of six target bacteria: Pseudomonas aeruginosa, Klebsiella spp., Stenotrophomonas maltophilia, Escherichia coli, Staphylococcus aureus, or Achromobacter xylosoxidans.

The study will enroll up to 30 participants across three U.S. clinical sites. Eligible subjects will receive a 7-day course of IV antibiotics prescribed by their clinical team, along with a pathogen-specific four-phage cocktail administered twice daily through a peripherally inserted central catheter (PICC). The phage cocktails are prepared under GMP conditions and have demonstrated lytic activity against clinical isolates of each target pathogen.

The primary endpoint is to evaluate the safety and tolerability of the combined phage-antibiotic therapy by monitoring adverse events (AEs), serious adverse events (SAEs), and events of special interest (ESIs). Secondary endpoints include changes in bacterial load in sputum (colony counts and qPCR), changes in lung function (spirometry and oscillometry), and patient-reported quality of life measures. An exploratory endpoint includes characterizing the pharmacokinetic profile of IV phage therapy in serum and sputum.

Initial doses of phage will be administered under direct clinical observation to monitor for immediate reactions. If well-tolerated, subsequent doses may be self-administered at home. Follow-up assessments will be conducted up to 28 days post-treatment, with additional safety monitoring extending up to 217 days. The trial is not designed to support regulatory approval but to generate essential safety and feasibility data to guide future efficacy trials in this high-need patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Confirmed diagnosis of cystic fibrosis.
* Sputum culture within 24 months and at screening showing at least one of the following: Pseudomonas aeruginosa, Klebsiella spp., Stenotrophomonas maltophilia, Escherichia coli, Staphylococcus aureus, or Achromobacter xylosoxidans.
* Percent predicted FEV₁ ≥ 40% (GLI).
* If ppFEV₁ > 40%, must have ≥ 1 pulmonary exacerbation per year requiring IV antibiotics or radiographic evidence of severe disease.
* Prior successful home IV antibiotic therapy within 5 years (may be waived by investigator).
* Available phage cocktail with lytic activity against the participant's pathogen.

Oxygen saturation > 88% on room air after rest. Able to provide written informed consent.

Exclusion Criteria:

* Untreated or uncontrolled mycobacterial or fungal airway infection.
* History of Clostridioides difficile without a negative test within 3 months. Concerning exotoxin, virulence, or resistance genes in the bacterial isolate (per investigator).
* Mixed-species bacterial infection at screening.
* Participation in another interventional trial within 30 days.
* Allergy or hypersensitivity to study materials.
* Pregnancy, planned pregnancy, or breastfeeding.
* Any condition or abnormality that, in the investigator's judgment, makes participation unsafe or may interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of combined IV antibiotic and bacteriophage therapy assessed by the number, type, severity, and relatedness of adverse events (AEs), serious adverse events (SAEs), and events of special interest (ESIs) | Baseline (Day -14 to Day 1) through Day 28 ± 5
  Safety will be assessed by the number, type, severity, and relatedness of adverse events (AEs), serious adverse events (SAEs), and events of special interest (ESIs) during and following the 7-day treatment period, in accordance with CTCAE criteria. Monitoring will occur from the initiation of the study drug through the 28-day follow-up period.

SECONDARY OUTCOMES:
Microbiological activity of combined IV antibiotic and bacteriophage therapy | Baseline (Day -14 to Day 1) through Day 28 ± 5
  Assessed by changes in bacterial burden in expectorated sputum samples, measured by quantitative culture (CFU/mL) and qPCR for the target pathogen. A response is defined as a ≥0.5 log reduction in bacterial load from baseline.
Microbiological Response: Sputum Bacterial Load (Quantitative Culture) measured by quantitative culture | From the first dose through 28 days after the last dose of study treatment
  Change in Sputum Bacterial Load (Quantitative Culture) measured by quantitative culture.
  Time Frame: Baseline to Day 36 Unit of Measure: CFU/mL
Change in Lung Function (FEV₁ Percent Predicted) measured by percent predicted forced expiratory volume in one second (FEV₁ % predicted). | Baseline to Day 36
  Change in Lung Function (FEV₁ Percent Predicted) measured by percent predicted forced expiratory volume in one second (FEV₁ % predicted).
  Unit of Measure: Percent predicted
Change in Respiratory Symptoms Using the Cystic Fibrosis Respiratory Symptom Diary - Chronic Respiratory Infection Symptom Score (Cystic Fibrosis Respiratory Symptom Diary-CRISS) | Baseline to Day 36
  Change in Respiratory Symptoms Using the Cystic Fibrosis Respiratory Symptom Diary - Chronic Respiratory Infection Symptom Score (Cystic Fibrosis Respiratory Symptom Diary-CRISS). Scores range from 0 (no symptoms) to 100 (most severe symptoms). Unit of Measure: Units on a 0-100 scale